CLINICAL TRIAL: NCT02040909
Title: Optimizing Propofol Dosing for (Preterm) Newborn Infants That Need Endotracheal Intubation
Acronym: NEOPROP2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: interim results concluded no added value of additional inclusion
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Maxima Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Stichting Nuts Ohra (Other)
Responsible Party: Principal Investigator, Sinno H.P. Simons, Dr.S.H.P. Simons, pediatrician-neonatologist, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20132312; 2013-005572-17 (EudraCT Number); 90713494 (Other Grant/Funding Number: ZonMW); 1201-020 (Other Grant/Funding Number: fondsNutsOhra)
Record Dates: First submitted 2013-12-23; First posted 2014-01-20 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia Intubation Complication; Premature Birth of Newborn; Other Preterm Infants; Propofol Overdose
Keywords: sedation; quality of intubation; hypotension; pharmacodynamics; pharmacokinetics
MeSH Terms: conditions — Premature Birth; Hypotension | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Experimental): A predetermined propofol dose is used in every 5 consecutive patients per age group. Starting dose is 1.0 mg/kg. Dose is increased or decreased with 0.5 mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol, an anesthetic agent, is used to sedate the patients before endotracheal intubation. The propofol starting dose in all age groups will be 1.0 mg propofol/kg. After 5 patients per age group the next dose will be determined. Dose will be increased or decreased with 0.5 mg/kg for the next 5 patients. The study will be continued untill an adequate dose, that results in adequate sedation, good intubation conditions without hypotension, is determined. That dose will be valideted in another 5 patients per age group.
  Other Names: Diprivan

SUMMARY:
Newborns admitted to an intensive care unit often require artificial ventilation. For that purpose an endotracheal tube needs to be placed into the trachea, a procedure named endotracheal intubation. The newborns need to be sedated to keep them comfortable, to stop moving and to relax in order to enable the success of the procedure. For this sedation an anesthetic agent named propofol is often used. The used dose of propofol has not been properly studied and as a consequence patients are under- or over -sedated and propofol leads to side effects such as hypotension.

The current study aims to find the most appropriate dose of propofol for newborns of different gestational ages and of different post-natal ages. We will use propofol in different doses and after each 5 included patients per age group we will analyze whether the dose needs to be increased or decreased. The effect of the propofol will be extensively monitored and we will study the level of sedation, the quality of intubation, the stability of the patient en the occurrence of side effects.

At the end we aim to have appropriate guidelines for propofol doses in newborns of all ages.

DETAILED DESCRIPTION:
Rationale: Propofol, a rapidly acting anaesthetic agent, is currently used unlicensed in the clinical care of (preterm) neonates as sedative for endotracheal intubation. Neonates receive the same propofol doses per kg bodyweight, independent of their developmental stage (gestational age, postnatal age), morbidity, co-medication, etc. This is related to a high failure rate of intubation attempts and leads to hypotension in around 40 percent of patients. Propofol research in newborn infants is on the recently published priority drug research list of the European Medicines Agency (EMA). Propofol metabolism and elimination (PK: pharmacokinetics) as well as propofol effects (PD: pharmacodynamics) highly depend on the stage of development and on the genetic make-up of a patient. This study is based on the hypotheses that currently used single doses of propofol for newborn infants can be optimized and that this will improve the quality of sedation and increase the safety of the patients.

Objective: To determine effective and safe age specific propofol dosing guidelines for neonates of different age groups (both gestational age and postnatal age). Secondary objective is to determine a new age specific PK/PD (pharmacokinetic/pharmacodynamic), including a specific propofol genotype (pharmacogenetic analyses) that enables much better prediction of the effects and side-effects of propofol.

Study design: Prospective single dose optimizing and dose validation study

Study population: Neonates admitted at the Neonatal Intensive Care Unit (gestational age 24 - 42 weeks, post natal age < 28 days divided into 8 different age groups) that need (semi-)elective endotracheal intubation.

Intervention (if applicable): Adapted propofol dose. Starting dose is dependent on effects of previously included patients. Dose is increased in case of insufficient sedation. Intubation is started only after sedation level is adequate (titration with additional propofol is possible because propofol is very fast acting)

Main study parameters/endpoints: Primary outcome is the appropriate dose of propofol in 8 different age groups. Optimized propofol doses need to be related with adequate sedation, good quality of intubation conditions and no short term side effects. Secondary endpoints include further evaluation of cerebral perfusion, stress levels and short and long term outcome of the included patients. The incorporation of PK data and genotype of patients is used to make a prediction model for future patients that includes various important cofactors, related to effects and side effects of propofol. Physiological and behavioural responses of the newborns are further explored to find the most reliable and validate neonatal sedation score for intubations.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Propofol is used as a standard of care for sedation before intubation in newborn infants. Drug metabolism, drug transporters and drug receptors are not yet well developed in (preterm) newborn infants. Therefore PK/PD is very much dependent on the developmental stage of the newborn infant and though changes with age. This study can therefore not be done in another patient group (for instance older patients or healthy volunteers).

Internationally used propofol starting doses in newborns vary between 1.0 to 2.5 mg/kg and are repeated if necessary. The current study will start with propofol doses of 1.0 mg/kg in every age group. If the study starting dose is insufficient, the patient will receive additional propofol doses (1.0 mg/kg) until adequate sedation is acquired. No patient will be intubated before adequate sedation is reached. This is possible because propofol is very fast acting (1-2 minutes).

If the starting dose turns out to be insufficient in 5 patients per group it will be increased in the following patients of that group. The effect of an initial propofol dose is tested to find the optimal propofol doses for neonates in different developmental stages. The study will be continued until the appropriate dose for each age group is determined. The appropriate doses are re-used in another 5 patients per age group to validate the predetermined doses. Safety is monitored very intensively and if hypotension occurs this is immediately treated. The patient will benefit from this intensive safety monitoring, because side-effects will be detected earlier and can be more effectively treated.

Included patients will be monitored with non-invasive techniques (videotaping, cranial ultrasound, aEEG, NIRS) next to the standard intensive care monitoring of physiological parameters.

Blood samples will only be collected from indwelling arterial lines or during routine blood sampling because of normal patients care. An amount of 1.7 ml blood (0.5 ml for DNA analyses, 2 times 0.6 ml for propofol PK analyses) is taken if possible. Two saliva samples for cortisol analyses will be collected.

ELIGIBILITY:
Inclusion Criteria:

All neonates admitted to the two participating intensive care units:

* Less than 28 days postnatal age
* Who need endotracheal intubation

Exclusion Criteria:

Patients with:

* Major congenital anomalies or neurological disorders,
* Neonates with an abnormal upper airway,
* Those receiving continuous sedatives or opioids, and
* Those whose mothers received sedatives or opioids before or during delivery will be excluded during the first 2 days of life.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
adequate propofol dose | 24 hours
  Adequate propofol doses are determined by 3 co-primary outcome variables:
  * Adequate sedation
  * Optimal intubation conditions
  * No hypotension or other severe side effects

SECONDARY OUTCOMES:
Determine a valid sedation assessment scale | 24 hours
  To develop a validated and useful sedation assessment instrument for (preterm) newborns during endotracheal intubation. For this aim validated pain assessment instruments (COMFORTneo, neonatal Pain And Sedation Scale, Premature Infant Pain Profile and Neonatal Infant Pain Scale will be compared with an available sedation score by the use of videotapes. Furthermore we aim to determine the relationship between these pain and sedation scores with the patients stress level as measured by cortisol levels.
to determine an age specific propofol PK/PD model | 24 hours
  Pharmacodynamic data of propofol are explored (duration of intubation, duration of sedation, time of side effect, recovery of spontaneous breathing). We will analyze propofol concentrations in a pharmacokinetic model and integrate pharmacodynamic data (level of sedation, side effects) and covariates (age, weight, morbidity, etc). We aim to determine effective propofol concentrations and concentrations that might result in side-effects.
aEEG / NIRS | 24 hours
  -To further explore dose and age-related hemodynamic effects of propofol. Next to blood pressure and heart rate cerebral oxygenation and continuous amplitude-integrated EEG (aEEG) will be monitored. After the intubation procedure, when the patient is still sedated the cerebral perfusion is measured using cerebral Doppler sonography. In this way we aim to determine the effects of propofol on cerebral perfusion. Risk factors for hypotension and cerebral hypoperfusion are determined.

OTHER OUTCOMES:
Propofol polymorphisms on effect and metabolizing enzymes | 1 year
  To further explain expected inter-individual variability in propofol concentrations and effects by adding genotypic variability to the PK/PD model. Polymorphisms in genes encoding propofol metabolizing enzymes (UGT 1A9 and Cytochrome P450 2B6) and GABA (gamma-aminobutyric acid) receptors will be analysed in the patients DNA

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam van Weissenbruch, MD PhD, Study Director — VU Medical Center Amsterdam
Locations (3):
- Netherlands (3):
  - VU Medical Center, Amsterdam
  - Erasmus MC Sophia Children's Hospital, Rotterdam
  - Maxima Medisch Centrum, Veldhoven